CLINICAL TRIAL: NCT05131165
Title: INcentives and ReMINDers to Improve Long-term Medication Adherence
Acronym: INMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mildmay Uganda Limited (Other); Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH122331 (NIH); R34MH122331 (NIH)
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS
Keywords: ART Adherence; Reminders; Behavioral Economics; Viral Suppression; Long-term Adherence; Routines; Habit Formation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled trial with two intervention arms and a control group, that will receive intervention for three months with follow-on assessment for six months after the intervention period ends.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will be blinded to treatment assignment of study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This arm will receive care as usual, including the adherence support mechanisms that are part of usual care practices. At recruitment participant will be explained the importance of pill-taking. All participants (including in the control group) will receive a leaflet containing detailed information on how to establish healthy pill-taking routines. Finally, clinic staff will counsel participants on how to select an already regularly routine behavior that occurs at roughly the same time each day that forms the basis of their implementation plan.
- Intervention group receiving messages (Messages Group) (Experimental): Participants will receive the same information as those in the Control Group, but in addition, receive the "Daily Text Message" Intervention.
  Interventions: Behavioral: Daily Text Messages
- Intervention group receiving messages and incentives (Incentives Group) (Experimental): Participants will receive the same information as the Control group. Additionally, they will receive the "Daily Text Message Intervention" and will be eligible for prize drawings.
  Interventions: Behavioral: Daily Text Messages; Behavioral: Incentivization based on timely ART adherence

INTERVENTIONS:
Behavioral: Daily Text Messages — Participants will receive daily text message reminders to use their routine behavior to trigger medication adherence.
  Arms: Intervention group receiving messages (Messages Group); Intervention group receiving messages and incentives (Incentives Group)
Behavioral: Incentivization based on timely ART adherence — Participants will be eligible to draw a prize if they take their medication within +/- one hour of the stated existing routine to which pill-taking is anchored on at least 70% of days between recruitment and the 3-month study visit.
  Arms: Intervention group receiving messages and incentives (Incentives Group)

SUMMARY:
The study will test the feasibility and acceptability of using text messages and behavioral economics-based incentives to support anchoring Anti-Retroviral Therapy (ART) adherence to an existing routine in order to improve long-term ART medication adherence. The intervention phase of the three-phased study will constitute the pilot RCT. A sample of 150 clients who have initiated ART in the preceding three months will be randomized to either usual care (C = 50) or one of the two INMIND intervention groups (daily text message reminders with or without incentives) for three months (T1 = 50; T2=50). Subsequently, behavioral persistence will be evaluated for six months post-intervention. Assessments will be conducted at baseline, month 3, and month 9. The primary outcomes are 1) electronically measured mean medication adherence during the intervention and 2) six months post intervention, along with 3) timeliness of medication adherence during the intervention and 4) six months post-intervention.

DETAILED DESCRIPTION:
Adherence of Anti-Retroviral Therapy (ART) among HIV-infected patients initiating treatment (treatment initiators) in Sub-Saharan Africa has remained low, even though the number of treatment initiators has increased in recent years. Lack of retention in care and low adherence in the first year of ART treatment are substantial barriers to virologic suppression. The current R34 study tests a novel approach for improving long-term ART adherence among treatment initiators by turning adherence into a behavioral routine. This is done in two ways: 1) anchoring ART adherence to an existing routine, and 2) providing more immediate rewards and increasing the salience through reminder messages. Insights from behavioral economics suggest that such an intervention may be particularly effective for people with present bias (those who have a tendency to give in to short-term temptation at the cost of more long-term benefits) and lack of salience (where over time, the choice of target behavior is overshadowed by more pressing needs of daily life) which have been found to be prevalent among people living with chronic medical conditions from past studies.

The intervention will be tested through a pilot RCT, wherein 150 adult clients will be randomly assigned to three groups. The first intervention group would receive daily text messages that reinforce routine formation information provided to all participants (across the three groups). The second intervention group will receive the text messages, and additionally be eligible for a prize drawing based on timely ART adherence, at each monthly clinic visit. The control group will receive care as usual, consisting of routine formation information as well as adherence counseling. The intervention will last three months, with a six-month post-intervention follow up period. All participants will receive MEMS caps to record adherence, and will complete assessments over nine months (baseline, post-intervention, and six months post-intervention).

The Specific Aim of the intervention phase of the study is to test the preliminary effectiveness of the intervention, including the relative effectiveness of the two different implementation approaches. This is preceded by the formative phase, with the Specific Aim of developing the intervention parameters. The intervention phase is succeeded by the adaptation phase, whose Specific Aim is to collect data in preparation for a subsequent R01 application.

ELIGIBILITY:
Inclusion Criteria:

* Male and female clients age 18 and older.
* Started ART at Mildmay or another clinic within the preceding three months but have since been receiving care at Mildmay.
* Able to speak and understand either English or Luganda.
* Have their own cell phone or have consistent access to someone else's phone.
* Willing to receive daily text messages for the 3 months of intervention duration.
* Willing and able to use the MEMS caps distributed for adherence verification for the duration of the study.

Exclusion Criteria:

* Not mentally fit to consent.
* Language other than Luganda or English.
* Not willing to consistently use the MEMS caps device for adherence measurement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Linnemayr, Ph.D., Principal Investigator — RAND
Locations (1):
- Mildmay Uganda Limited, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data collected in the execution of the aims described in the application will be shared in the form of journal publications. Following publication of the main paper(s) for this study and the grant end-date, the RAND Human Subjects Protection Committee will be consulted about how to securely make data publicly available in the form of an electronic database for researchers who successfully complete a registration process (described below). Any shared data will be de-identified and will not contain any direct identifiers or indirect identifiers (that could identify participants by inference). No qualitative data will be shared, as such data would be difficult to de-identify given that participants will be telling their own experiences and thus could be identified by inference. Documentation of shared data will be provided in the form of a codebook in which each variable name and response options are defined.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be decided after consultation with the RAND Human Subjects Protection Committee.
Access Criteria: Access will be allowed post-registration, wherein accessing individuals will need to completed a data sharing agreement that outlines the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. The data sharing agreement will include a commitment to using the data only for research purposes, a commitment to securing the data using appropriate computer technology, and a commitment to destroying or returning the data after analyses are completed. Users must submit brief proposals regarding intended use of the data; the study team will determine the scientific soundness of the proposal as part of the decision for the researcher to be able to access the public use dataset.

REFERENCES:
- [Background] Ruppar TM, Russell CL. Medication adherence in successful kidney transplant recipients. Prog Transplant. 2009 Jun;19(2):167-72. doi: 10.1177/152692480901900211. PMID 19588667
- [Background] Phillips LA, Gardner B. Habitual exercise instigation (vs. execution) predicts healthy adults' exercise frequency. Health Psychol. 2016 Jan;35(1):69-77. doi: 10.1037/hea0000249. Epub 2015 Jul 6. PMID 26148187
- [Background] Lally P, Wardle J, Gardner B. Experiences of habit formation: a qualitative study. Psychol Health Med. 2011 Aug;16(4):484-9. doi: 10.1080/13548506.2011.555774. PMID 21749245
- [Background] Stecher C, Mukasa B, Linnemayr S. Uncovering a behavioral strategy for establishing new habits: Evidence from incentives for medication adherence in Uganda. J Health Econ. 2021 May;77:102443. doi: 10.1016/j.jhealeco.2021.102443. Epub 2021 Mar 16. PMID 33831632
- [Background] Stecher C, Linnemayr S. Promoting antiretroviral therapy adherence habits: a synthesis of economic and psychological theories of habit formation. AIDS. 2021 Apr 1;35(5):711-716. doi: 10.1097/QAD.0000000000002792. No abstract available. PMID 33306553
- [Background] Jennings Mayo-Wilson L, Devoto B, Coleman J, Mukasa B, Shelton A, MacCarthy S, Saya U, Chemusto H, Linnemayr S. Habit formation in support of antiretroviral medication adherence in clinic-enrolled HIV-infected adults: a qualitative assessment using free-listing and unstructured interviewing in Kampala, Uganda. AIDS Res Ther. 2020 Jun 8;17(1):30. doi: 10.1186/s12981-020-00283-2. PMID 32513192
- [Background] Linnemayr S, Stecher C. Behavioral Economics Matters for HIV Research: The Impact of Behavioral Biases on Adherence to Antiretrovirals (ARVs). AIDS Behav. 2015 Nov;19(11):2069-75. doi: 10.1007/s10461-015-1076-0. PMID 25987190
- [Background] Linnemayr S, Stecher C, Mukasa B. Behavioral economic incentives to improve adherence to antiretroviral medication. AIDS. 2017 Mar 13;31(5):719-726. doi: 10.1097/QAD.0000000000001387. PMID 28225450
- [Background] Linnemayr S, Huang H, Luoto J, Kambugu A, Thirumurthy H, Haberer JE, Wagner G, Mukasa B. Text Messaging for Improving Antiretroviral Therapy Adherence: No Effects After 1 Year in a Randomized Controlled Trial Among Adolescents and Young Adults. Am J Public Health. 2017 Dec;107(12):1944-1950. doi: 10.2105/AJPH.2017.304089. Epub 2017 Oct 19. PMID 29048966
- [Derived] Linnemayr S, Odiit M, Mukasa B, Ghai I, Stecher C. INcentives and ReMINDers to Improve Long-Term Medication Adherence (INMIND): impact of a pilot randomized controlled trial in a large HIV clinic in Uganda. J Int AIDS Soc. 2024 Jun;27(6):e26306. doi: 10.1002/jia2.26306. PMID 38923298
- [Derived] Stecher C, Ghai I, Lunkuse L, Wabukala P, Odiit M, Nakanwagi A, Linnemayr S. Incentives and Reminders to Improve Long-term Medication Adherence (INMIND): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 31;11(10):e42216. doi: 10.2196/42216. PMID 36315224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a randomized, parallel controlled trial, a sample of 166 participants who met the inclusion criteria were recruited at Mildmay Uganda between October, 2021 and April, 2022. Participants were excluded if a) they did not own an phone, b) they started ARTs > 3 months prior to enrollment, c) they were not at Mildmay general or planned to transfer our during the study period, d) could not offer informed consent, or e) could not commit to study activities
Pre-assignment Details: After recruitment but prior to random assignment and baseline assessment, enrolled participants were given a MEMS cap to screen for non-use (recorded adherence < 30% over a month). Of 166 enrolled, 3 participants were excluded due to MEMS non-use, 3 did not return for baseline, and 1 withdrew consent at baseline, leaving 159 participants to randomize. Of these, 2 in the control group and 1 in the Messages group withdrew consent after baseline and thus their data are not reported in the flow.
Groups:
- Control: This arm will receive care as usual, including the adherence support mechanisms that are part of usual care practices. At recruitment participant will be explained the importance of pill-taking. All participants (including in the control group) will receive a leaflet containing detailed information on how to establish healthy medication-taking routines. Finally, clinic staff will counsel participants on how to select an already established routine behavior that occurs at roughly the same time each day that forms the basis of their implementation plan.
- Intervention Group Receiving Messages (Messages Group): Participants will receive the same information as those in the Control Group, but in addition, receive the "Daily Text Message" Intervention for the first three months after baseline.
  Daily Text Messages: Participants will receive daily text message reminders to use their routine behavior to trigger medication adherence.
- Intervention Group Receiving Messages and Incentives (Incentives Group): Participants will receive the same information as the Control group. Additionally, they will receive the "Daily Text Message Intervention" and will be eligible for "incentivization based on timely ART adherence" for the first three months after baseline.
  Daily Text Messages: Participants will receive daily text message reminders to use their routine behavior to trigger medication adherence.
  Incentivization based on timely ART adherence: Participants will be eligible to draw a prize if they take their medication within +/- one hour of the stated existing routine to which pill-taking is anchored on at least 70% of days between recruitment and the 3-month study visit.
Period: Overall Study
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Started | 50 | 51 | 58
Completed Month-3 Visits (Completed the month-3 visits, which included a survey, and the final administration of conditional incentives for the Incentives group) | 44 | 46 | 54
Completed (Completed the final study visit, scheduled at around 9 months after baseline.) | 45 | 46 | 50
Not Completed | 5 | 5 | 8
Not completed — Death | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 5
Not completed — Transferred out of clinic | 1 | 0 | 3
Not completed — Dropped out | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group) | Total
Number analyzed (Participants) | 49 | 49 | 58 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.06 (8.33) | 33.57 (8.90) | 34.84 (11.34) | 33.9 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 40 | 103
  Male | 17 | 18 | 18 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 49 | 49 | 58 | 156
Number of children [Mean (Standard Deviation); unit: children] | 2.37 (2.13) | 2.94 (3.27) | 2.70 (2.16) | 2.67 (2.55)
Monthly income [Mean (Standard Deviation); unit: USD] | 59.20 (119.29) | 78.02 (81.71) | 72.95 (116.55) | 70.10 (107.26)
Travel to clinic: Cost [Mean (Standard Deviation); unit: USD] | 3.79 (3.72) | 3.52 (3.49) | 3.33 (2.39) | 3.53 (3.20)
Travel to clinic: Time (Hrs) [Mean (Standard Deviation); unit: hours] | 1.14 (0.62) | 1.19 (0.91) | 1.41 (2.59) | 1.25 (1.68)
% disclosed HIV status [Count of Participants; unit: Participants] | 43 | 40 | 47 | 130
% primary education or less [Count of Participants; unit: Participants] | 21 | 24 | 25 | 70
% married (or partnered) [Count of Participants; unit: Participants] | 31 | 23 | 33 | 87
% employed at baseline [Count of Participants; unit: Participants] | 35 | 40 | 46 | 121
% food insecure [Count of Participants; unit: Participants] — Calculated based on the Food Insecurity Experience Scale (FIES): participants with a food insecurity score >3 were considered to have high food insecurity
  Participants | 11 | 13 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Pills Taken as Prescribed Over the Intervention Period (Baseline - Month 3)
Description: MEMS-data was collected continuously over the course of the three-month intervention period allowing us to investigate mean adherence. Only one of the ART medications was used to calculate the primary adherence variable (# of actual bottle openings / # of prescribed bottle openings).
Time Frame: Three months
Population: Includes all enrolled participants with at least one day's adherence data from the MEMS cap between baseline and month 3 visits (n = 155).
Measure: Least Squares Mean (Standard Error); unit: Proportion of pills taken as prescribed
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Number analyzed (Participants) | 49 | 49 | 57
Proportion of pills taken as prescribed | 0.860 (0.027) | 0.916 (0.030) | 0.914 (0.028)
Statistical Analysis 1: Comparison: Control vs Intervention Group Receiving Messages (Messages Group); The analyses utilized control as the reference group, and thus, the values reported include control mean and standard error as the reference value (derived from an ordinary least squared regression without controls). The results for the intervention groups are derived from the multiple regression model that controlled for other participant characteristics, including demographics, intrinsic motivation and habit strength at baseline; Test type: Superiority; p = 0.056, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05
Statistical Analysis 2: Comparison: Control vs Intervention Group Receiving Messages and Incentives (Incentives Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.062, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05

2. Primary Outcome: Proportion of Pills Taken as Prescribed Over the Post-intervention Period (Months 4-9)
Description: MEMS-data was collected continuously over the course of the six-month post intervention period allowing for the investigation of post-intervention mean adherence. Only one of the ART medications was used to calculate the primary adherence variable (# of actual bottle openings / # of prescribed bottle openings).
Time Frame: Six months post-intervention
Population: Includes all enrolled participants with at least one day's adherence data from the MEMS cap between months 4-9 (n = 135).
Measure: Least Squares Mean (Standard Error); unit: Proportion of pills taken as prescribed
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Number analyzed (Participants) | 43 | 42 | 50
Proportion of pills taken as prescribed | 0.800 (0.029) | 0.842 (0.038) | 0.835 (0.032)
Statistical Analysis 1: Comparison: Control vs Intervention Group Receiving Messages (Messages Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.364, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05
Statistical Analysis 2: Comparison: Control vs Intervention Group Receiving Messages and Incentives (Incentives Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.409, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05

3. Primary Outcome: Proportion of Pills Taken Within +/- 1 Hour of the Anchor Time Over the Intervention Period (Baseline - Month 3)
Description: A novel measure of routine adherence (that it is explicitly based on the temporal pattern of pill-taking), calculated as the fraction of scheduled pills taken within a one-hour window around the typical time that participants report completing their existing routine behavior that anchors their pill-taking, was calculated. This measure provides an objective way for determining behavioral automaticity of pill-taking.
Time Frame: Three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Proportion of pills taken in time window
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Number analyzed (Participants) | 49 | 49 | 57
Proportion of pills taken in time window | 0.685 (0.041) | 0.755 (0.05) | 0.81 (0.05)
Statistical Analysis 1: Comparison: Control vs Intervention Group Receiving Messages (Messages Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.158, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05
Statistical Analysis 2: Comparison: Control vs Intervention Group Receiving Messages and Incentives (Incentives Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.017, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05

4. Primary Outcome: Proportion of Pills Taken Within +/- 1 Hour of the Anchor Time Over the Post-Intervention Period (Months 4-9)
Description: This measure would be calculated as a fraction of scheduled pills taken within a one-hour window around the typical time that participants report completing their existing routine behavior that anchors their pill-taking, for all visits made post-intervention.
Time Frame: Six months post-intervention
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Proportion of pills taken in time window
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Number analyzed (Participants) | 43 | 42 | 50
Proportion of pills taken in time window | 0.546 (0.047) | 0.573 (0.066) | 0.680 (0.064)
Statistical Analysis 1: Comparison: Control vs Intervention Group Receiving Messages (Messages Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.654, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05
Statistical Analysis 2: Comparison: Control vs Intervention Group Receiving Messages and Incentives (Incentives Group); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.035, ANCOVA — A priori threshold for statistical significance (alpha) = 0.05

5. Secondary Outcome: Retention in Care
Description: Retention in care was measured as the fraction of participants recruited who are still active clients at the clinic at month 9.
Time Frame: Month 9
Population: All participants that consented to participate and were randomized to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Number analyzed (Participants) | 50 | 51 | 58
Participants | 48 | 50 | 57

6. Secondary Outcome: Change in Viral Suppression Status
Description: HIV RNA (viral load) was the secondary outcome measure. For each participant, viral loads taken just prior to baseline and viral loads taken just after month-9 were compared; if participant was virally suppressed (with < 200 copies of HIV per millilitre (mL) of blood) at baseline, but had a viral load of >= 200 copies/mL after month-9, then the indicator was assigned "-1"; if there was no change in viral suppression status (i.e., if participant either had >= 200 copies of virus/mL at baseline and month-9 OR if participant had < 200 copies/mL at baseline and month-9), then the indicator was assigned "0". If, however, the participant's viral load went from >= 200 copies/mL at baseline to < 200 copies/mL after month-9, then the indicator was assigned "1".
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: indicator score
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
Number analyzed (Participants) | 33 | 37 | 41
indicator score | 0.03 (0.175) | 0 (0.039) | 0 (0.035)
Statistical Analysis 1: Comparison: Control vs Intervention Group Receiving Messages (Messages Group); The analyses compared the change in viral suppression status of the participants from baseline to month 9. For each participant, we derived the change in viral suppression status by subtracting two binary variables - one indicating whether the participant was virally suppressed at baseline (based on their chart records from around 3 months prior to baseline) and the other indicating whether the participant was virally suppressed at around month 9 of the study; Test type: Superiority; p = 0.5468, t-test, 2 sided
Statistical Analysis 2: Comparison: Control vs Intervention Group Receiving Messages and Incentives (Incentives Group); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.5255, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 10 months (recruitment - month 9)
Description: We used the same definition for all cause mortality as the ClinicalTrials.gov definition. Given that our intervention was behavioral in nature, targeting participants that were already in treatment for HIV, we did not expect any participant to be at risk for All-Cause Mortality.
Arm/Group | Control | Intervention Group Receiving Messages (Messages Group) | Intervention Group Receiving Messages and Incentives (Incentives Group)
All-Cause Mortality (participants affected / at risk) | 1/51 | 1/50 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/58
Other Adverse Events (participants affected / at risk) | 0/51 | 0/50 | 0/58

LIMITATIONS AND CAVEATS:
Limitations consist of our statistical analysis being based on a small pilot study that was not powered for all outcomes. Also, the intervention took place in a single HIV clinic in Uganda, but we believe the intervention site (and hence our results) to be fairly representative of many urban clinics in sub-Saharan Africa.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT05131165/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05131165/ICF_000.pdf